CLINICAL TRIAL: NCT05226520
Title: Effect of 6-week Probiotic Supplementation on Stress-related Parameters in Healthy Adults With Different Levels of Stress
Brief Title: Psychophysiological Effects of Probiotic Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2004NRC
Record Dates: First submitted 2021-12-06; First posted 2022-02-07 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Mild to Moderate Levels of Stress

STUDY DESIGN:
Intervention Model Description: Exploratory, randomized, placebo-controlled, 2-arms, double-blinded, parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unique coding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic NCC3001 (Experimental): Sachets of NCC3001 and excipient (maltodextrin) to be administered orally every day for 6 weeks
  Interventions: Dietary Supplement: Experimental probiotic product
- Matched Placebo Comparator (Placebo Comparator): Sachets of matching placebo containing maltodextrin, yeast extract, cystein HCl and pea flour to be administered orally every day for 6 weeks
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Dietary Supplement: Experimental probiotic product — Probiotic supplementation
  Arms: Probiotic NCC3001
Other: Placebo comparator — Placebo
  Arms: Matched Placebo Comparator

SUMMARY:
This is a pilot exploratory study to investigate the effects of a probiotic Bifidobacterium longum NCC3001 intake on physiological and psychophysiological parameters related to stress in healthy individuals with mild to moderate stress level.

DETAILED DESCRIPTION:
The purpose of the study is to explore the effects of a probiotic Bifidobacterium longum NCC3001 intake on physiological and psychophysiological parameters related to stress in healthy individuals with mild to moderate stress level.

The objectives is three:

* Measure the effects of a 6-week supplementation with NCC3001 on psychological and physiological parameters in response to an acute experimental stress;
* Measure the effects of a 6-week supplementation with NCC3001 on chronic stress level, gastro-intestinal symptoms and sleep quality;
* Explore changes in the profiles of biological parameters associated with ingestion of NCC3001; including changes in hormones, neurotransmitters, circulating immune and microbiome-derived molecules and changes in the microbiome itself

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign the informed consent
2. Healthy adult men and/or women aged 25 to 65 years old
3. Mild to moderate stress, defined as a score in the range of 15 to 25 on the validated Depression, Anxiety and Stress Scale (DASS-42)
4. Proficiency in French and/or English
5. Normal visual acuity and hearing with or without correction (self-reported)
6. BMI in the range of 18.5 to 29.9 kg/m2

Exclusion Criteria:

1. Diagnosed food allergies
2. Currently participating or having recently participated in a clinical study with products potentially interfering with the results as judged by the investigator
3. Organic gastrointestinal pathology other than benign polyps, diverticulosis, hemorrhoids
4. Chronic or recurrent diarrhea with spontaneous bowel movements more often than 2 times daily
5. Concurrent diagnosed systemic chronic disease (e.g., endocrine, cardiovascular, metabolic, liver, celiac)
6. Willing to avoid the consumption of probiotic-containing products (including yogurts containing probiotics) i.e. any commercially available product specified as containing Lactobacillus, Bifidobacteria, Streptococcus or Saccharomyces for the 2 weeks prior to randomization visit
7. Willing to avoid the use of antibiotics in the 4 weeks prior to randomization visit
8. Adherence to an overly unbalanced diet such as vegan, paleo, ketogenic, low carbohydrate, raw diets
9. Conditions that may affect mood

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol level | Before the stressor (time-point -20 minutes) and after the stressor (time-point +0 min, time-point +5 min, time-point +10 min, time-point +20 min, time-point +30 min, time-point +40 min) at both baseline and after 6 weeks of treatment
  Salivary cortisol levels (nmol/L) before and after stressor

SECONDARY OUTCOMES:
Cortisol level from waking saliva samples | Baseline and after 6 weeks treatment
  Cortisol level (nmol/L) from waking saliva samples collected 0, 15, 30, 45, 60 min after waking
Mean heart rate variability | Baseline and after 6 weeks treatment
  Mean heart rate variability in the time (ms) measured continuously before, during and after the stressor by means of a portable a computer-based data acquisition system from Biopac, Inc
Heart frequency | Baseline and after 6 weeks treatment
  Heart frequency (Hz) measured continuously before, during and after the stressor by means of a portable a computer-based data acquisition system from Biopac, Inc
Mean skin conductance level | Baseline and after 6 weeks treatment
  Mean skin conductance level (SCL, kΩ) measured continuously before, during and after the stressor by means of a portable a computer-based data acquisition system from Biopac, Inc
Self-reported measures before and after the stressor (PANAS) | Baseline and after 6 weeks treatment
  Positive and negative affect scores (1-50) computed with the Positive and Negative Affect Schedule (PANAS)
Self-reported measures before and after the stressor (STAI-6) | Baseline and after 6 weeks treatment
  Likert scores (1-4) for 6 mood dimensions: calm, tense, upset, relaxed, content, worry from the State Trait Anxiety Inventory 6-item short form (STAI-6)
Self-reported measures before, during and after the stressor (VAS) | Baseline and after 6 weeks treatment
  VAS scores in mm (0-100) for subjective perception of the stress induction
Self-reported endpoints from standard questionnaires (PSS) | Baseline and after 6 weeks treatment
  Perceived stress score (0-56) computed from the Perceived Stress Scale (PSS)
Self-reported endpoints from standard questionnaires (HADs) | Baseline and after 6 weeks treatment
  Scores (0-21) of depression and anxiety computed from the Hospital Anxiety and Depression scale (HADs)
Self-reported endpoints from standard questionnaires (GSRS) | Baseline and after 6 weeks treatment
  Scores from the Gastrointestinal Symptom-Rating Scale (GSRS): scores range from 1 to 7 and higher scores represent more discomfort
Self-reported endpoints from standard questionnaires (Pittsburgh Sleep Quality) | Baseline and after 6 weeks treatment
  Sleep quality score from the Pittsburgh Sleep Quality Index questionnaire (score 0-21: the lower, the better sleep quality)
Probiotic in feces | Baseline and after 6 weeks treatment
  Probiotic quantity in feces (genome copy number / million 16S copy number)
Microbiome related metabolites in stool, blood and urine | Baseline and after 6 weeks treatment
  Microbiome related metabolites in stool, blood and urine

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Macé, Study Director — Nestlé Institute of Health Science
Locations (1):
- Nestlé Research, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
No plan